CLINICAL TRIAL: NCT04318470
Title: Using Metagenomic Next-generation Sequencing to Identify Microbial DNA in Maternal Plasma in Cases of Preterm Premature Rupture of Membranes
Brief Title: Identification of Microbial DNA in Maternal Plasma After PPROM
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 10-00505-JD
Record Dates: First submitted 2020-03-10; First posted 2020-03-24 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Preterm Rupture of Membranes
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PPROM: Preterm premature rupture of membranes between 16 0/7 and 33 6/7 weeks gestation
  Interventions: Diagnostic Test: mNGS
- Healthy controls: Gestational-age-matched controls without preterm premature rupture of membranes or other pregnancy complications
  Interventions: Diagnostic Test: mNGS

INTERVENTIONS:
Diagnostic Test: mNGS — Metagenomic next generation sequencing for microbial DNA

SUMMARY:
This study evaluates the use of metagenomic next generation sequencing in identifying microbial DNA in plasma samples of patients with preterm premature rupture of membranes.

DETAILED DESCRIPTION:
Although preterm premature rupture of membranes (PPROM) occurs in only 3% of pregnancies, it accounts for 30% of preterm births (PTB) and is associated with serious maternal and neonatal morbidity. An important factor in the underlying pathophysiology of PPROM and subsequent PTB is subclinical infection, which promotes a cascade of events that contribute to synthesis of prostaglandins, release of proinflammatory cytokines, infiltration of neutrophils, and activation of metalloproteases. Over time, enhanced activity of these infectious and inflammatory pathways contributes to the development of spontaneous labor and/or overt intraamniotic infection (IAI). Unfortunately, the majority of patients with PPROM do not manifest signs and symptoms of infection that are detectable by clinical examination, laboratory evaluation, and traditional microdiagnostic tests, and attempting to predict length of latency period and/or timing of delivery remains a clinical challenge. We propose the use of metagenomic next-generation sequencing (mNGS) to identify microbial DNA in maternal plasma following PPROM. We hypothesize that the presence and abundance of microbial DNA is associated with a shorter latency period and that an increase in the abundance of microbial DNA precedes delivery.

ELIGIBILITY:
Inclusion Criteria:

* For PPROM group, preterm premature rupture of membranes between 16 0/7 and 33 6/7 weeks of gestation
* For control group, healthy pregnancy with no evidence of preterm premature rupture of membranes or other major complications

Exclusion Criteria:

* Maternal age < 18 years
* Major fetal congenital malformation

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant patients with preterm premature rupture of membranes and gestational-age-matched controls
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Length of latency | From study enrollment to date of delivery, up to 24 weeks
  Time between PPROM and delivery

SECONDARY OUTCOMES:
Maternal infectious morbidity | From study enrollment to date of delivery, up to 30 weeks
  Composite of fever, intrauterine infection, sepsis, postpartum endometritis, surgical site infection, and administration of antibiotics
Neonatal infectious morbidity | From neonatal birth to neonatal hospital discharge, up to 1 year
  Composite of fever, sepsis, administration of antibiotics, and need for blood/urine/cerebrospinal fluid (CSF) cultures
Histopathological signs of infection | At time of placental delivery
  Histopathological signs of infection on routine post-delivery examination of placenta, membranes, and umbilical cord
Perinatal demise | From study enrollment to 28 days of life
  Composite of intrauterine fetal demise and neonatal demise
Admission to neonatal intensive care unit (NICU) | From neonatal birth to neonatal hospital discharge, up to 1 year
NICU length of stay | From neonatal birth to neonatal hospital discharge, up to 1 year
Neonatal need for supplemental oxygen | From neonatal birth to neonatal hospital discharge, up to 1 year
Respiratory distress syndrome | From neonatal birth to neonatal hospital discharge, up to 1 year
Necrotizing enterocolitis | From neonatal birth to neonatal hospital discharge, up to 1 year
Intraventricular hemorrhage | From neonatal birth to neonatal hospital discharge, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nasim C Sobhani, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No